CLINICAL TRIAL: NCT03043924
Title: Functional Study of the Hypothalamus in High-resolution Magnetic Resonance Imaging (MRI) in Women With Polycystic Ovary Syndrome (PCOS): a Comparative Study
Brief Title: Functional Study of the Hypothalamus in Magnetic Resonance Imaging (MRI) in Polycystic Ovary Syndrome (PCOS)
Acronym: MRI-PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2016_22; 2016-A01391-50 (Other: ID-RCB Number, ANSM)
Record Dates: First submitted 2017-01-31; First posted 2017-02-06 (Estimated); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Polycystic Ovary Syndrome
Keywords: hypothalamus; Diffusion Magnetic Resonance Imaging; Magnetic Resonance Spectroscopy
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Cyproterone Acetate; Estradiol; Levonorgestrel; Ethinyl Estradiol; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCOS women (Other): 26 PCOS women who receive consultation for hyperandrogenism needing treatment with Cyproterone Acetate + estradiol will be recruited.
  Interventions: Drug: Cyproterone Acetate + estradiol
- Healthy volunteers (Other): 26 Healthy volunteers subjects who receive consultation contemplating oral contraceptives (Levonorgestrel, Ethinyl Estradiol 0.1-0.02Mg Oral Tablet ) will be recruited.
  Interventions: Drug: Levonorgestrel, Ethinyl Estradiol 0.1-0.02Mg Oral Tablet

INTERVENTIONS:
Drug: Cyproterone Acetate + estradiol — PCOS will receive:
  50mg cyproterone acetate (Androcur®) in combination with p.o. 2mg estradiol daily
  Other Names: Androcur, Provames
  Arms: PCOS women
Drug: Levonorgestrel, Ethinyl Estradiol 0.1-0.02Mg Oral Tablet — Healthy volunteers receive combined oral contraceptive (COC) consisting 0.02 mg ethinylestradiol and 0.1mg of progestins (Leeloo Gé®)
  Other Names: Leeloo Gé®
  Arms: Healthy volunteers

SUMMARY:
The aim to evaluate whether activation of the hypothalamic-pituitary-gonadal axis in PCOS is associated with transient microstructural and metabolic changes in the female hypothalamus using MRI approaches to assess water diffusion and measure proton magnetic resonance spectra.

ELIGIBILITY:
Inclusion Criteria:

For all subjects

* Aged from 19 to 30 years
* Body mass index : 18-25
* Informed consent before inclusion
* Do not smoke the 3 days before the MRI

For Healthy volunteers subjects :

* Regular cycles (between 25 and 35 days) AND ovulatory.
* No signs of hyperandrogenism.
* Subjects desirous of taking oral contraceptives (estrogen/progestin combination).
* For the realization of the 2nd MRI: to be during the 3rd month of a treatment well followed by oestro-progestative monophasic minidose to 0,02mg of Ethinyl-oestradiol / 0,1mg Levonorgestrel.

PCOS women:

* PCOS defined by Rotterdam criteria
* Needing a treatment with cyproterone acetate
* To carry out the 2nd MRI: to be in progress during the 3rd month of a treatment well followed by 50 mg of Cyproterone acetate in association with 2mg / day of natural estradiol.

Exclusion Criteria:

* Hormone treatment within 3 months prior to inclusion (including birth control pill )
* On-going pregnancy (determined before each MRI scan visit)
* Claustrophobia
* Any metal or foreign implants (e.g., aneurysm clips, ear implants, heart pacemakers or defibrillators)
* Diabetes or known dysthyroidism.
* Current substance abuse (including smoking more than 5 cigarettes/day; determined using drug screening at the screening visit)
* Pregnancy or breastfeeding the last 3 months.
* Practice of intense physical exercise (ex jogging> 10km) the day before the MRI.
* Person incapable of consenting, or enjoying legal protection (guardianship / curatorship).
* Unability to understand the treatment protocol

Ages: 19 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Change in the Apparent Diffusion Coefficient (ADC) | Baseline and 3 months after treatment start
  The change in the ADC will be analyzed in healthy volunteers and PCOS women before starting the oral contraceptives, and next during the third sequence of treatment.

SECONDARY OUTCOMES:
Change in the metabolite concentrations | Baseline and 3 months after treatment start
  The change in the metabolite concentrations will be analyzed in the two groups before starting the oral contraceptives, and next during the third sequence of treatment.
Correlation coefficient (Spearman or Pearson) between the ADC and serum hormonal levels (FSH,luteinizing hormone,oestradiol, AMH) | Baseline and 3 months after treatment start
  The correlation between ADC and hormonal levels in the two groups will be analysed before starting the contraceptive treatment and during the third processing sequence.
Correlation coefficient (Spearman or Pearson) between the metabolite concentrations and serum hormonal levels (FSH, luteinizing hormone, oestradiol, AMH) | Baseline and 3 months after treatment start
  The correlation between metabolite concentrations and hormonal levels in the two groups will be analysed before starting the contraceptive treatment and during the third processing sequence.
Plasma GnRH concentration before and after treatment (PCOS patient and control group) | Baseline and 3 months after treatment start
Correlation between brain metabolite concentrations and plasma GnRH concentration before and after contraception. | Baseline and 3 months after treatment start

CONTACTS AND LOCATIONS:
Overall Officials: Didier Dewailly, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Jeanne de Flandres, CHU, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Barbotin AL, Mimouni NEH, Kuchcinski G, Lopes R, Viard R, Rasika S, Mazur D, Silva MSB, Simon V, Boursier A, Pruvo JP, Yu Q, Candlish M, Boehm U, Bello FD, Medana C, Pigny P, Dewailly D, Prevot V, Catteau-Jonard S, Giacobini P. Hypothalamic neuroglial plasticity is regulated by anti-Mullerian hormone and disrupted in polycystic ovary syndrome. EBioMedicine. 2023 Apr;90:104535. doi: 10.1016/j.ebiom.2023.104535. Epub 2023 Mar 29. PMID 37001236